CLINICAL TRIAL: NCT01401920
Title: The Influence of Passive Leg Elevation on the Cross-sectional Area of the Internal Jugular Vein in Infants or Young Children Undergoing Open Heart Surgery
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Chung Su Kim, Professor, Samsung Medical Center
Other Study IDs: 2011-05-093
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Infants or Children Undergoing Open Heart Surgery
Keywords: internal jugular vein cannulation; cross-sectional area; passive leg elevation; trendelenburg position; open heart surgery
MeSH Terms: interventions — Head-Down Tilt; Control Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients undergoing open heart surgery: small infant or children patients undergoing open heart surgery
  Interventions: Other: leg elevation; Other: Trendelenburg position; Other: Trendelenburg position + passive leg elevation; Other: control group

INTERVENTIONS:
Other: leg elevation — bilateral passive leg elevation for 30 seconds
Other: Trendelenburg position — Trendelenburg position (15 degrees) for 30 seconds
Other: Trendelenburg position + passive leg elevation — Trendelenburg position + passive leg elevation
Other: control group — supine position without passive leg elevation or trendelenburg position

SUMMARY:
The trendelenburg position is usually applied to increase the cross-sectional area of the IJV. However, trendelenburg position requires a tilt table to place the head in the down position. Trendelenburg position could also increase intracranial pressure. Passive leg elevation redistributes more blood from the lower extremity into the central veins and is proved to increase the cross-sectional area of IJV in adults. However, the effect of leg elevation on the cross-sectional area of IJV in small infants and children has not been evaluated.

The investigators evaluated the effect of passive leg elevation on the cross-sectional area of IJV in subjects undergoing open heart surgery for congenital anomaly.

DETAILED DESCRIPTION:
Internal jugular vein (IJV) cannulation is essential for open heart surgery of small infants and children for transfusion or inotropics infusion. The trendelenburg position is usually applied to increase the cross-sectional area of the IJV.

However, trendelenburg position requires a tilt table to place the head in the down position. Trendelenburg position could also increase intracranial pressure. Passive leg elevation redistributes more blood from the lower extremity into the central veins and is proved to increase the cross-sectional area of IJV in adults. However, the effect of leg elevation on the cross-sectional area of IJV in small infants and children has not been evaluated. Furthermore, the children undergoing open heart surgery due to cardiac anomaly have an altered hemodynamics and often congested right heart. Therefore, the response of passive leg elevation may be different from that of normal heart physiology. Therefore, we evaluated the effect of passive leg elevation on the cross-sectional area of IJV in subjects undergoing open heart surgery for congenital anomaly.

ELIGIBILITY:
Inclusion Criteria:

* infants or children under 5 yrs undergoing elective open heart surgery for congenital anomaly for study period

Exclusion Criteria:

* previous history of internal jugular vein cannulation
* concurrent pulmonary disease that can influence the hemodynamics of right heart
* increased intracranial pressure
* hemodynamic unstability

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants or children undergoing open heart surgery for congenital anomaly for study period
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Cross-sectional area of internal jugular vein | one time measurement 10 min before jugular vein cannulation
  Cross-sectional area of internal jugular vein measured on the ultrasonographic image with planimetry method

SECONDARY OUTCOMES:
Transverse diameter of internal jugular vein | only one time measurements 10 min before internal jugular vein cannulation
  Transverse diameter of internal jugular vein measured on the ultrasonographic image
horizontal diameter of internal jugular vein | only one time measurements 10 min before jugular vein cannulation
  horizontal diameter of internal jugular vein measured on the ultrasonographic image
skin to internal jugular vein depth | one time measurement 10 min before jugular vein cannulation
  skin to internal jugular vein depth measured on the ultrasonographic image

CONTACTS AND LOCATIONS:
Overall Officials: Chung Su Kim, M.D.,Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea